CLINICAL TRIAL: NCT05112861
Title: A 3-month Study to Compare the Safety of ONS-5010 in Vials Versus PFS in Subjects With Visual Impairment Due to Retinal Disorders, NORSE SEVEN
Brief Title: A 3-month Study to Compare the Safety of ONS-5010 in Vials Versus Pre-filled Syringe in Subjects With Visual Impairment Due to Retinal Disorders
Acronym: NORSE SEVEN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Outlook Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONS-5010-007
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Age-Related Macular Degeneration; Neovascular Age-related Macular Degeneration; Wet Macular Degeneration; BRVO - Branch Retinal Vein Occlusion; Diabetic Macular Edema
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Retinal Vein Occlusion | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Biological: bevacizumab (Experimental)
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — 1.25 mg, intravitreal injection
  Other Names: ONS-5010

SUMMARY:
The study will compare the safety of ophthalmic bevacizumab in vials versus pre-filled syringes in subjects diagnosed with a retinal condition that would benefit from treatment with intravitreal injection of bevacizumab, including: exudative age-related macular degeneration, diabetic macular edema, or branch retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Active clinical diagnosis and OCT confirmation of one of the following retinal disorders: exudative age-related macular degeneration (AMD), diabetic macular edema (DME), or branch retinal vein occlusion (BRVO) and, in the opinion of the Investigator, requires treatment with an anti-VEGF therapy

Exclusion Criteria:

* Previous use of approved anti-VEGF or Avastin® within 4 weeks preceding randomization
* Previous use of Beovu®
* Macular edema due to something other than exudative AMD, DME or BRVO, in the study eye
* History of inadequate response to previous intravitreal anti-VEGF therapy
* History of any intraocular or periocular corticosteroid injection or implant, in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1-month preceding randomization
* Any concurrent intraocular condition in the study eye that may require medical or surgical intervention or contribute to vision loss during the study period
* Active intraocular inflammation in the study eye
* Current vitreous hemorrhage in the study eye
* Polypoidal choroidal vasculopathy (PCV) in the study eye
* History of idiopathic, infectious or autoimmune-associated uveitis in either eye
* Current ocular or periocular infection, such as conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with anti-glaucoma medication)
* Premenopausal women not using adequate contraception
* Current treatment for active systemic infection
* Known allergy to any component of the study drug , not amenable to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Frequency and incidence of treatment-emergent adverse events following intravitreal injections of ONS-5010 in vials or PFS | 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Site, Springfield, Illinois
  - Clinical Site, Hagerstown, Maryland
  - Clinical Site, Chambersburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No